CLINICAL TRIAL: NCT02662712
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, First-in-human Study of Orally Administered JNJ-56136379 to Evaluate Safety, Tolerability and Pharmacokinetics After Single Ascending Doses and One Multiple Dose Regimen in Healthy Subjects (Part I), and After Multiple Dose Regimens in Subjects With Chronic Hepatitis B (Part II)
Brief Title: A Study of Orally Administered JNJ-56136379 to Evaluate Safety, Tolerability and Pharmacokinetics After Single Ascending Doses and One Multiple Dose Regimen in Healthy Participants (Part I), and After Multiple Dose Regimens in Participants With Chronic Hepatitis B (Part II)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CR108092; 56136379HPB1001 (Other: Janssen Sciences Ireland UC); 2015-003724-30 (EudraCT Number)
Record Dates: First submitted 2015-12-02; First posted 2016-01-25 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Hepatitis, Chronic
Keywords: Healthy; Hepatitis, Chronic; JNJ-56136379; Placebo
MeSH Terms: conditions — Hepatitis, Chronic | interventions — JNJ-56136379

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Device: No

ARMS (3):
- Part 1: Single Dose Escalation (Experimental): The single dose escalation phase of the study will consist of 6 dosing sessions (Sessions I to VI) evaluated in 2 panels (Panels 1 and 2). The dose of JNJ-56136379 will be consecutively escalated over 5 levels, alternating between the 2 panels. Panel 1 will receive 3 single doses (SD1, SD3 and SD3fed) in Sessions I, III and V, respectively. Panel 2 will receive 3 single doses (SD2, SD4 and SD5) in Sessions II, IV and VI, respectively. There will be a washout period of at least 14 days between consecutive JNJ-56136379/placebo dosing in each individual participant.
  Interventions: Drug: JNJ-56136379; Drug: Placebo
- Part 1: Multiple dose session (Experimental): After completion of the fifth single dose session another panel of healthy participant (panel 3) receive multiple doses of JNJ-56136379 at one dose level (MDx) or placebo for 12 or 19 consecutive days (Session VII) in fed or fasted conditions.
  Interventions: Drug: JNJ-56136379; Drug: Placebo
- Part 2: Multiple dose escalation (Experimental): Multiple dose levels will be given in Panel 4 in Session VIII (European sites), Sessions IX and X (European and/or Asian sites) Session XI (Asian sites) for 28 consecutive days in fed conditions. Optional Sessions A-B-C (Panel 4) used for further dose evaluations at European and/or Asian sites. Per session, participants will receive JNJ 56136379 or placebo. Dose progression to the next multiple dose level may be adapted based on the emerging safety and PK outcome of the previous dosing levels.
  Interventions: Drug: JNJ-56136379; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-56136379 — JNJ-56136379 oral tablets will be given in Part 1 (single dose escalation and multiple dose session) and Part 2 (multiple dose escalation).
Drug: Placebo — Matching placebo to JNJ-56136379 will be given in Part 1 (single dose escalation and multiple dose session) and Part 2 (multiple dose escalation).

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and safety data including serious and other adverse events, physical examinations, vital signs, 12-lead electrocardiograms (ECGs) and clinical laboratory results (including biochemistry, hematology, and urine).

DETAILED DESCRIPTION:
Part 1: This is a first-in-human (FIH), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), randomized (study medication assigned to participants by chance), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study. Part 1 includes healthy adult participants, divided into 3 panels (Panel 1, 2 and 3) and in Part 2 adult Chronic Hepatitis B Participants will be included, in Sessions VIII to XI and Optional Sessions A-B-C (Panel 4). The study will consists of screening phase (part 1: [less than or equal to <=28 days before the first intake of study drug; part 2: [<=56 to greater than or equal to {>=} 20 days before the first intake of study drug), Treatment Phase (multiple dose phase in part 1: Day -1 up to 12 or 19 days; part 2: up to 4 weeks) and Follow up Phase (part 1: 30-35 days after last study drug intake or after dropout; part 2: up to week 8 after actual end of study drug treatment). Participants' safety will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* For Part II, a female participant must be either of a) Non-childbearing potential defined as: 1) Postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level (greater than (>)40 international unit per milliliter (IU/L) or milli-international units per milliliter (mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient, or 2) Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy, or b) Childbearing potential and practicing sexual abstinence or a highly effective method of contraception from screening onwards and agree to continue to use the same method of contraception throughout study treatment and for at least 90 days after the last dose of study drug (or longer, if dictated by local regulation)
* Female participants should have a negative serum pregnancy test at screening
* Healthy Participants: Participants must have a body mass index (BMI; weight in kg divided by the square of height in meters) of 18.0 to 30.0 kilogram per square meter (kg/m2), extremes included
* Chronic Hepatitis B Participants: Participants must have lack of advanced liver disease, ie, either: Metavir F0-F2 (or comparable histologic scoring system) as determined on a liver biopsy within one year of the screening visit; a result based on specific radiologic liver disease staging modalities (eg, Fibroscan, AFRI, magnetic resonance imaging [MRI]-Elastography) compatible with Metavir F0-F2 within 6 months of the screening visit
* Chronic Hepatitis B Participants: Participants must have HBV DNA of greater than or equal [>=] 2,000 international unit per milliliter (IU/mL) at screening
* Chronic Hepatitis B Participants: Participants must be aged between 18 years to 65 years, have a body mass index (BMI; weight in kg divided by the square of height in meters) of 18.0 to 35.0 kilogram per square meter (kg/m^2), extremes included

Exclusion Criteria:

* Healthy Participants: Participants with a past history of cardiac arrhythmias (example, extrasystolic, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Healthy Participants: Female participants who are breastfeeding at screening
* Healthy Participants: Participants with current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* Chronic Hepatitis B Participants: Participants with current HCV infection (confirmed by HCV antibody or HCV RNA) or hepatitis delta virus (HDV) infection (confirmed by HDV antibody) at screening
* Chronic Hepatitis B Participants: Participants with positivity of anti-HBs antibodies
* Chronic Hepatitis B Participants: Participants with a past history of cardiac arrhythmias (eg, extrasystolic, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Chronic Hepatitis B Participants: Female participants who are breastfeeding at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Part 1 Single Ascending Dose and Multiple Dose : Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events | Until the last study-related activity (30-35 days after last dosing)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 2: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events | Up to Week 12
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 1 Single Ascending Dose and Multiple Dose : Number of Participants With Abnormal Physical Examinations | 30-35 days after last study drug intake or after dropout
  Physical examinations (including body weight measurement and skin examination) will be performed.
Part 2: Number of Participants With Abnormal Physical Examinations | Up to Week 8
  Physical examinations (including body weight measurement and skin examination) will be performed.
Part 1 Single Ascending Dose and Multiple Dose : Number of Participants With Abnormal Vital Signs | 30-35 days after last study drug intake or after dropout
  Vital signs (Supine Blood Pressure [SBP], Diastolic Blood Pressure [DBP] pulse rate: supine and standing) will be performed.
Part 2: Number of Participants With Abnormal Vital Signs | Up to Week 8
  Vital signs (SBP, DBP pulse rate: supine and standing) will be performed.
Part 1 Single Ascending Dose and Multiple Dose : Number of Participants With Clinically Significant Laboratory Findings | 30-35 days after last study drug intake or after dropout
  The laboratory abnormalities will be determined according to the criteria specified in the World Health Organization (WHO) Toxicity Grading Scale and in accordance with the normal ranges of the clinical laboratory.
Part 2: Number of Participants With Clinically Significant Laboratory Findings | Up to Week 8
  The laboratory abnormalities will be determined according to the criteria specified in the World Health Organization (WHO) Toxicity Grading Scale and in accordance with the normal ranges of the clinical laboratory.
Part 1: Maximum Observed Plasma Concentration (Cmax) After Single Dose Administration | Pre-dose, 0.5 hour (hr), 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hr post-dose on Day 1
  Cmax is the Maximum observed plasma concentration.
Part 1: Maximum Observed Plasma Concentration (Cmax) After Multiple Dose Administration | Pre-dose, 0.5 hr, 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hr Day 1; post-dose on Day 12
  Cmax is the Maximum observed plasma concentration.
Part 2: Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 8, 12 hr post-dose on Day 1; post-dose on Day 28
  Cmax is the Maximum observed plasma concentration.
Part 1: Area Under the Curve From Time 0 to the Time of the Last Measurable Concentration (AUClast) After Single Dose Administration | Pre-dose, 0.5 hour (hr), 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hr post-dose on Day 1
  AUClast is the area under the curve from time 0 to the time of the last measurable Concentration.
Part 2: Area Under the Curve From Time 0 to the Time of the Last Measurable Concentration (AUClast) | Pre-dose, 8, 12 hr post-dose on Day 1; post-dose on Day 28
  AUClast is the area under the curve from time 0 to the time of the last measurable Concentration.
Part 1: Area Under the Curve From Time 0 to Infinity (AUC infinity) After Single Dose Administration | Pre-dose, 0.5 hour (hr), 1, 1.5, 2, 3, 4, 6, 8, 12 and 16 hr post-dose on Day 1
  AUC infinity is the area under the curve from time 0 to infinity.
Part 2: Area Under the Curve From Time 0 to Infinity (AUC infinity) | Pre-dose, 8, 12 hr post-dose on Day 1; post-dose on Day 28
  AUC infinity is the area under the curve from time 0 to infinity.

SECONDARY OUTCOMES:
Part 2: Change From Baseline in Mean Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) | Up to week 12
  HBV DNA will be quantified using an in vitro nucleic acid amplification test for the quantification of HBV DNA.
Part 2: Maximum Decrease in HBV DNA (Baseline-subtracted Mean) | Up to week 12
  HBV DNA will be quantified using an in vitro nucleic acid amplification test for the quantification of HBV DNA.
Part 2: Changes in Hepatitis B Surface Antigen (HBsAg) Levels | Up to week 12
  Quantitative HBsAg and levels will be determined from samples using standard serologic assays.
Part II: Percentage of Participants with Treatment Emerging Mutations | Up to week 12
  Treatment induced emerging mutations will be assessed by comparing the HBV genome sequence obtained at baseline with sequences obtained post-baseline.
Part II: Change From Baseline in HBV DNA (Antiviral Activity) in Chronic Hepatitis B (CHB) Participants with Sequence Variations in the HBV Genome | Up to week 12
  Sequence variations in the HBV genome will be assessed by sequencing of the viral genome. Antiviral activity will be assessed by measuring change from baseline in HBV DNA concentration using in vitro nucleic acid amplification test for the quantification of HBV DNA and compared between participants with and without HBV sequence variations.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (27):
- Belgium (4):
  - Brussels
  - Edegem
  - Mechelen
  - Merksem
- Sofia, Bulgaria
- France (4):
  - Clichy
  - La Tronche
  - Lyon
  - Paris
- Tbilisi, Georgia
- Germany (3):
  - Essen
  - Hanover
  - Wiesbaden
- Kuala Lumpur, Malaysia
- Chisinau, Moldova
- Romania (2):
  - Bucharest
  - Timișoara
- Spain (5):
  - Barcelona
  - Madrid
  - Santander
  - Seville
  - Valencia
- Taiwan (5):
  - Kaohsiung City
  - Keelung
  - Taichung
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Zoulim F, Lenz O, Vandenbossche JJ, Talloen W, Verbinnen T, Moscalu I, Streinu-Cercel A, Bourgeois S, Buti M, Crespo J, Manuel Pascasio J, Sarrazin C, Vanwolleghem T, Shukla U, Fry J, Yogaratnam JZ. JNJ-56136379, an HBV Capsid Assembly Modulator, Is Well-Tolerated and Has Antiviral Activity in a Phase 1 Study of Patients With Chronic Infection. Gastroenterology. 2020 Aug;159(2):521-533.e9. doi: 10.1053/j.gastro.2020.04.036. Epub 2020 Apr 25. PMID 32343960
- [Derived] Vandenbossche J, Jessner W, van den Boer M, Biewenga J, Berke JM, Talloen W, De Zwart L, Snoeys J, Yogaratnam J. Pharmacokinetics, Safety and Tolerability of JNJ-56136379, a Novel Hepatitis B Virus Capsid Assembly Modulator, in Healthy Subjects. Adv Ther. 2019 Sep;36(9):2450-2462. doi: 10.1007/s12325-019-01017-1. Epub 2019 Jul 2. PMID 31267367